CLINICAL TRIAL: NCT00988923
Title: Hyperthermia As A Conservative Treatment For Carpal Tunnel Syndrome. A Randomized "Sham" Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Giuseppina Frasca-Physical Medicine and Rehabilitation Department, Catholic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1198/07
Record Dates: First submitted 2009-06-12; First posted 2009-10-02 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group a: Hyperthermia (HT) (Experimental): HT were treated for 20 minutes per session, a total of 8 sessions with device;
  Interventions: Other: group A: HYPERTHERMIA
- group b: No intervention (No Intervention): device was switched in off, only bolus was active
  Interventions: Other: No intervention

INTERVENTIONS:
Other: group A: HYPERTHERMIA — All patients were treated for 8 sessions, twice a week, for a total of 4 weeks of treatment. All patients were evaluated at baseline (T0) and after 4 weeks (T1). The first two sessions were sham-treatment for both groups
  Other Names: HT produce heating.
  Arms: group a: Hyperthermia (HT)
Other: No intervention — the intervention tool was switched in off, only bolus was activated
  Other Names: simulated intervention
  Arms: group b: No intervention

SUMMARY:
The purpose of this study is to verify the short-term effects of hyperthermia (HT) in pain relief and in functional impairment in patients affected by mild to moderate idiopathic carpal tunnel syndrome.

A single blind randomized sham-controlled trial was performed. A 23 patients were affected by idiopathic CTS, 11 of them were affected by bilateral CTS.

the intervention consists of Hyperthermia device treatment, treated for 20 minutes per session, a total of 8 sessions. Primary outcome is pain (Visual analogic scale).

DETAILED DESCRIPTION:
Background: Non-surgical treatment is generally administered to patients with mild to moderate symptoms. Many of these treatments used heat modality. Hyperthermia is a relative recent device which produces deep heating.

Objective: The purpose of this study is to verify the short-term effects of hyperthermia (HT) in pain relief and in functional impairment in patients affected by mild to moderate idiopathic carpal tunnel syndrome.

Design: A double blind randomized sham-controlled trial. Setting: Outpatient physical therapy, institutional clinic. Participants: 23 patients were affected by idiopathic CTS, 11 of them were affected by bilateral CTS.

Intervention: Hyperthermia (HT) device treatment, treated for 20 minutes per session, a total of 8 sessions.

Measurement: Primary outcome is pain (Visual analogic scale). Secondary outcomes were self-reported pain intensity and physical functioning questionnaire (Levine/Boston), ultrasonographic (median nerve cross sectional area mnCSA) and neurophysiological data.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral or unilateral mild to moderate carpal tunnel syndrome confirmed by clinical and neurophysiological tests, with no indication to surgical intervention.
* All patients were grouped into first, second and third classes according to Historic and Objective (Hi-Ob)15 scale of CTS and minimum, mild CTS according to the neurophysiological classification of Padua1

Exclusion Criteria:

* Secondary entrapment neuropathies (diabetes, systemic disease)
* Cancer, pregnancy
* Electroneurographic and clinical signs of axonal degeneration of the median nerve.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome is visual analogic scale for pain (VAS) | 4 weeks

SECONDARY OUTCOMES:
Secondary outcomes were self-reported pain intensity and physical functioning questionnaire (Levine/Boston), ultrasonographic (median nerve cross sectional area (mnCSA) and neurophysiological data | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppina Frasca, MD, Principal Investigator — Rehabilitation Department, Catholic University, Rome
Locations (1):
- Department of Physical Medicine and Rehabilitation,, Roma, Rome, Italy